CLINICAL TRIAL: NCT02157363
Title: POsitioning for Esophageal Cancer Resection - a Randomized Controlled TRIal (POETRI)
Brief Title: POsitioning for Esophageal Cancer Resection
Acronym: POETRI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor recruitment due to change of surgical technique
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TW-001
Record Dates: First submitted 2014-05-12; First posted 2014-06-06 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Patient Positioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Repositioning Group (Active Comparator): The patient is placed on a vacuum mattress in supine position for the abdominal part using a midline laparotomy. After completion of the abdominal part, the abdomen is closed and dressed in standard fashion and the patient is repositioned under full anesthesia is a left-lateral decubitus (LLD) position. After the thorax is sterile prepped and draped, a right dorso-lateral thoracotomy in the 4th to 6th intercostal space under preservation of body of the serratus muscle is performed.
  Interventions: Procedure: Repositioning
- Single positioning (Experimental): The patient is placed on a vacuum mattress and in a left-screwed supine position for the entire operative procedure. The pelvis and the lower extremities are placed at 0° rotation, whereas the torso is rotated leftwards to an angle of 45° (Fig. 1). The patient is prepped and draped from the shoulders to the inguinal region. A midline laparotomy is done for the abdominal part and the abdomen closed afterwards. For the thoracic part, the operating table is tilted about 30° to the left, and a right anterolateral thoracotomy is performed in the 4th to 6th intercostal space.
  Interventions: Procedure: Single positioning

INTERVENTIONS:
Procedure: Repositioning
  Arms: Repositioning Group
Procedure: Single positioning
  Arms: Single positioning

SUMMARY:
Open thoracoabdominal esophagectomy (TAE) is the standard curative treatment modality for resectable esophageal cancer. TAE can be achieved by positioning the patient in the supine position for the abdominal part and in a left-lateral decubitus (LLD) position for the thoracic part, or by performing both parts in a left-screwed supine position (LSS). Aim of the present study is to compare peri- and postoperative outcome variables after TAE for esophageal cancer in the two positions.

POETRI is designed as a single-center, randomized controlled trial with two parallel arms including patients with resectable esophageal cancer and type I cancers of the esophagogastric junction (AEG I). Exclusion criteria are inability to tolerate surgery or both types of positioning, inability to perform an intrathoracic anastomosis, non-malignant pathologies. The primary endpoint is operating time. Secondary endpoints are morbidity, lymph node yield, pulmonary function, pain control and wound healing assessed during a follow-up of 3 months.

POETRI is a single-center, randomized controlled trial to evaluate different positioning and thoracic access during radical open thoracoabdominal esophagectomy for patients with resectable esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, non-metastatic esophagus cancer (squamous or adenocarcinoma) or AEG I tumors requiring curative thoracoabdominal esophagectomy with intrathoracic anastomosis of a gastric tube immediately after diagnosis or after neoadjuvant treatment
* Patients are considered fit for surgery by a local interdisciplinary team of surgeons, medical oncologists and anesthesiologists (ECOG performance status of 0,1, or 2).
* Age ≥ 18 years
* Written informed consent

Exclusion Criteria:

* Preoperative established indication for colon interposition or cervical anastomosis
* Preoperative diagnosed tracheo-esophageal fistula
* History of right thoracotomy or prior lung surgery
* Physical inability of the described intraoperative patient positioning
* Non-malignant esophageal pathology or other malignancies except squamous or adenocarcinoma
* Planned laparoscopic or thoracoscopic surgical approach
* Patients not eligible for TAE (ASA ≥ 4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
operating time | The endpoint is assessed at the end of the operation (finishing of all wound dressings) on the day of operation.
  Operating time is defined from the start of patient positioning until final closing and dressing of all wounds.

CONTACTS AND LOCATIONS:
Overall Officials: Thilo Welsch, MD, Principal Investigator — Department of Surgery, University Hospital Dresden
Locations (1):
- Department of Surgery, University Hospital Dresden, Dresden, Germany